CLINICAL TRIAL: NCT04335370
Title: Pharmacokinetics of Polymyxin B in Adult Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Shijing Jia, Assistant Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00150013
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis; Polymyxin B
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CF lung disease receiving Polymyxin B (PMB): Participants receiving polymyxcin B as part of standard of care treatment for CF exacerbation will have blood drawn measure blood concentrations of PMB
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood samples will be collected from enrolled patients at 5 time points during a single dosing interval:
  1. Prior to start of infusion
  2. End of infusion
  3. One hour after end of infusion
  4. Three hours after end of infusion
  5. Eight hours after start of infusion

SUMMARY:
Cystic fibrosis (CF) pulmonary disease is a major cause of morbidity and mortality in CF patients and is punctuated by episodes of acute exacerbation that require antibiotic treatment. Pseudomonas aeruginosa is the predominant bacterial pathogen isolated in patients with acute exacerbations, and practice guidelines recommend combination antibiotics directed against this pathogen as initial therapy. Such therapy traditionally consists of an antipseudomonal beta-lactam with either an antipseudomonal fluoroquinolone or an aminoglycoside. With growing P. aeruginosa multi-drug resistance, more adult patients present with isolates resistant to these traditional options.

The polymyxins are a class of cyclic peptide antibiotics that exert bactericidal activity through binding to the lipopolysaccharide component of gram-negative bacterial membranes and include colistin and polymyxin B (PMB). In recent years, there is growing evidence of increased rates of acute kidney injury associated with colistin in critically ill patients. Additionally, population pharmacokinetic (PK) studies suggest that fixed drug dosing may yield an improved therapeutic index over the traditional weight-based dosing of this agent. Thus there is growing interest in use of PMB as an alternative in CF acute exacerbations but the optimal dosage regimen is not known.

This is a single-center, open-label, non-interventional study to characterize the pharmacokinetics and safety of fixed-dose PMB in adult patients with CF by measuring serum concentrations in patients receiving IV therapy as a part of routine care. This study will help to validate existing population PK models and allow for adjustment of patient specific covariates (i.e. weight, renal function) unique to adult patients with CF. The study will also monitor for nephrotoxicity and neurotoxicity to determine if PMB has an acceptable margin of safety in this patient population. This investigation is the first to prospectively validate the pharmacokinetics and toxicities of fixed-dose PMB in CF and will guide optimal use of this compound in the management of acute pulmonary exacerbations.

DETAILED DESCRIPTION:
This study initially planned to include "Change in forced expiratory volume in one second (FEV1)" and "Non-response to therapy" as secondary outcome measures. These outcome measures were removed, as the small number of participants prohibited collection of significant data beyond what was collected for the baseline measures.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. Diagnosis of CF.
3. Receiving polymyxin B in the course of routine care.

Exclusion Criteria:

1. Evidence of acute kidney injury during the 48 hours prior to and following initiation of PMB therapy.
2. Extracorporeal organ support (including ECMO, iHD, and CRRT).
3. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CF patients admitted to the University of Michigan hospitals requiring polymyxin B as part of clinical care
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Polymyxin B compartmental population pharmacokinetics model | From immediately prior to a dose of therapy through 8 hours after therapy, approximately 8 hours
  The population pharmacokinetics of polymyxin B will be modeled based on the observed polymyxin B1 and B2 concentrations in plasma from enrolled patients who receive at least 1 dose of polymyxin B

SECONDARY OUTCOMES:
Acute kidney injury | From 48 hours after first dose through 48 hours after end of therapy, approximately 7-21 days depending on the length of the prescribed therapy
  Frequency of acute kidney injury occurring between 48 hours after initiation of polymyxin B and 48 hours after end of therapy
Neurotoxicity | From initiation of first dose through end of therapy, approximately 7-21 days depending on the length of the prescribed therapy
  Frequency of neurotoxicities occurring during polymyxin B treatment as documented by the primary clinical team
Change in forced expiratory volume in one second (FEV1) | FEV1 at baseline to 7 days post treatment, approximately 14-90 days in total
  After completion of polymyxin B therapy as documented by the primary clinical team
Non-reponse to therapy | From initiation of therapy through end of therapy, approximately 7-21 days depending on prescribed length of therapy
  Proportion of subjects requiring a change to antibiotic therapy due to non-response as documented by the primary clinical team

CONTACTS AND LOCATIONS:
Overall Officials: Shijing Jia, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crass RL, Al Naimi T, Wen B, Souza E, Murray S, Pai MP, Jia S. Pharmacokinetics of Polymyxin B in Hospitalized Adults with Cystic Fibrosis. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0079221. doi: 10.1128/AAC.00792-21. Epub 2021 Jul 12. PMID 34252297

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT04335370/Prot_SAP_000.pdf